CLINICAL TRIAL: NCT03622177
Title: Role of the IL33/Amphiregulin Pathway as a Potential Therapeutic Target in HIV Infection : a Prospective Cross-sectional Observational Study
Brief Title: Role of the IL33/Amphiregulin Pathway as a Potential Therapeutic Target in HIV Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS EP65 AMVIH
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: HIV I Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV+
  Interventions: Procedure: biopsie; Biological: blood drawn
- HIV- STI+
  Interventions: Procedure: biopsie
- HIV- STI-
  Interventions: Procedure: biopsie

INTERVENTIONS:
Procedure: biopsie — Additional colorectal mucosal biopsies during rectoscopy or colonoscopy
Biological: blood drawn — Additional blood drawn by venepuncture
  Groups: HIV+

SUMMARY:
Interleukin33 organize local immune reactions, especially at epithelial barriers.

ST2 is the IL33 receptor. The sST2 rate is higher for patient living with HIV and is an independent predictable factor of mortality. Interleukin33 induce tissue Treg ST2+ lymphocytes proliferation and amphireguline production. Amphireguline is member of epithelial growth factors family, which contributes to tissue repair, and fibrose. Amphireguline also helps immunosuppressives functions. Targetting amphiregulin for people living with HIV who has poor restauration of LTCD4+ could be a future therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1: HIV-infected subjects

   * HIV-1 infection
   * Age ≥ 18 years old
   * CD4 count≥ 100/mm3
   * Receiving an active antiretroviral treatment (plasma HIV viral load ≤ 50 copies/ml)
   * Subjects needing an STI screening for routine care including rectal biopsy (independently of the current study protocol)

   NB : an additional inclusion criteria for the Group 1 will be defined after the "phase 0" which will define two levels of fibrosis (low / high)
2. Group 2: controls not infected with HIV needing a rectoscopy for an STI screening

   * HIV negative
   * Age ≥ 18 years old
   * Subjects needing an STI screening for routine care including rectal biopsy (independently of the current study protocol)
3. Group 3: controls not infected with HIV needing a colonoscopy

   * HIV negative
   * Age ≥ 18 years old
   * Subjects needing a colonoscopy with colorectal biopsy as part of routine care (independently of the current study protocol)

For the 3 groups:

Inclusion criteria

* Affiliated or beneficiary of a Social Security coverage
* Free, informed and written consent, signed by the participant and the investigator (at the latest on the day of pre-inclusion and before any examination carried out within the framework of the trial)

Exclusion Criteria for the 3 groups

* - HIV-2 infection or HIV-1 & HIV-2 co-infection
* Active infection or cancer
* Contraindication to rectal biopsies (coagulation disorders, anticoagulation therapy, anorectal surgery, inflammatory bowel disease, post-radial rectitis)
* Subject participating in another research evaluating other treatments with an exclusion period ongoing at the screening visit.
* Person under legal guardianship or deprived of liberty by a judicial or administrative decision.
* Pregnant or breastfeeding women
* Replicative HCV or HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people living with HIV compare to people who are not living with HIV :
  - people with high burden of STI / people without burden of STI
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Quantification of amphiregulin plasma levels | through study completion, an average of 1 year
  Quantification of amphiregulin plasma levels in HIV-infected subjects and correlation these levels with blood TCD4 cell count and clinical parameters (cardiac diastolic dysfunction, organ dysfunctions likely to be secondary to fibrosis phenomena) recorded in the CARDAMONE cohort.
Phenotypic characterization of gut Treg cells and CD8+ T lymphocytes (CTL) isolated from the intestinal mucosa | through study completion, an average of 1 year
Study of fibrosis markers in the intestinal mucosa | through study completion, an average of 1 year
In vitro functional analysis of amphiregulin from isolated CTL of the lamina propria | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Characterization of HIV reservoir of the digestive mucosa | through study completion, an average of 1 year
  (i) Analysis at the blood and digestive compartment (rectum) for different CD4 CD32a T lymphocyte populations, marker of the viral reservoir; (ii) Quantification HIV DNA and the HIV reservoir competent for replication from blood and gut
Determination of antiretroviral drugs levels in digestive tissue and in plasma and correlation between antiretroviral drugs levels and viral reservoir and lymphocyte phenotype | through study completion, an average of 1 year